CLINICAL TRIAL: NCT01921387
Title: A Phase I/II Study Evaluating Escalating Doses of 90Y-BC8-DOTA (Anti-CD45) Antibody Followed by BEAM Chemotherapy and Autologous Stem Cell Transplantation for High-Risk Lymphoid Malignancies
Brief Title: Radiolabeled Monoclonal Antibody and Combination Chemotherapy Before Stem Cell Transplant in Treating Patients With High-Risk Lymphoid Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ajay Gopal, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2728.00; NCI-2013-01378 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2728.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA044991 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2013-08-09; First posted 2013-08-13 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Hodgkin Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent T-Cell Non-Hodgkin Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Hodgkin Lymphoma; Refractory Mantle Cell Lymphoma; Refractory T-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Hodgkin Disease; Lymphoma, Mantle-Cell; Lymphoma, T-Cell | interventions — Carmustine; carmustine, poliferprosan 20 drug combination; Cytarabine; Etoposide; Melphalan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (90Y-BC8-DOTA, chemotherapy, PBSC) (Experimental): Patients receive yttrium Y 90 anti-CD45 monoclonal antibody BC8 IV on day -14. Patients also receive carmustine IV over 3 hours on day -7, etoposide IV over 2 hours BID on days -6 to -3, cytarabine IV over 4 hours BID on days -6 to -3, and melphalan IV over 30 minutes on day -2. Patients then undergo autologous PBSC transplant on day 0.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carmustine; Drug: Cytarabine; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Procedure: Peripheral Blood Stem Cell Transplantation; Radiation: Yttrium Y 90 Anti-CD45 Monoclonal Antibody BC8

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous PBSC transplant
  Other Names: autologous stem cell transplantation
Drug: Carmustine — Given IV
  Other Names: BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; Carmustin; Carmustinum; FDA 0345; Gliadel; N,N'-Bis(2-chloroethyl)-N-nitrosourea; Nitrourean; Nitrumon; SK 27702; SRI 1720; WR-139021
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo autologous PBSC transplant
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Radiation: Yttrium Y 90 Anti-CD45 Monoclonal Antibody BC8 — Given IV
  Other Names: 90Y Anti-CD45 MoAb BC8

SUMMARY:
This phase I/II trial studies the side effects and the best dose of radiolabeled monoclonal antibody when given together with combination chemotherapy before stem cell transplant and to see how well it works in treating patients with high-risk lymphoid malignancies. Radiolabeled monoclonal antibodies, such as yttrium Y 90 anti-CD45 monoclonal antibody BC8, can find cancer cells and carry cancer-killing substances to them without harming normal cells. Giving chemotherapy before a stem transplant stops the growth of cancer cells by stopping them from dividing or killing them. Stem cells collected from the patient's blood are then returned to the patient to replace the blood-forming cells that were destroyed by the radiolabeled monoclonal antibody and chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum-tolerated dose (MTD) of 90Y-BC8-DOTA (yttrium Y 90 anti-CD45 monoclonal antibody BC8) (anti-cluster of differentiation [CD] 45) that can be delivered prior to myeloablative carmustine, etoposide, cytarabine, and melphalan (BEAM) chemotherapy and autologous stem cell transplant (ASCT) for patients with high-risk B-non-Hodgkin lymphoma (NHL), T-NHL, and Hodgkin lymphoma (HL).

II. To evaluate the efficacy of 90Y-BC8-DOTA when administered at the estimated MTD prior to BEAM chemotherapy and ASCT for patients with high-risk B-NHL, T-NHL, and HL compared to historical controls treated with BEAM alone.

SECONDARY OBJECTIVES:

I. To describe the toxicity observed from the addition of 90Y-BC8-DOTA to BEAM.

II. To optimize the protein dose (Ab) to deliver a favorable biodistribution in the majority of patients.

III. To describe response rates and overall survival of patients with high-risk B-NHL, T-NHL, and HL following administration of 90Y-BC8-DOTA plus BEAM prior to ASCT.

IV. To describe the impact of rituximab concentrations, B-cell depletion, and disease burden on CD45 targeting.

V. To assess the correlation of lymphoma biomarkers with outcomes.

VI. To evaluate the effects of nodal-targeted irradiation by 90Y-BC8-DOTA on immune reconstitution following ASCT.

OUTLINE: This is a phase I, dose-escalation study of yttrium Y 90 anti-CD45 monoclonal antibody BC8 followed by a phase II study.

Patients receive yttrium Y 90 anti-CD45 monoclonal antibody BC8 intravenously (IV) on day -14. Patients also receive carmustine IV over 3 hours on day -7, etoposide IV over 2 hours twice daily (BID) on days -6 to -3, cytarabine IV over 4 hours BID on days -6 to -3, and melphalan IV over 30 minutes on day -2. Patients then undergo autologous peripheral blood stem cell (PBSC) transplant on day 0.

After completion of study treatment, patients are followed up at 3, 6, and 12 months and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of B-NHL, T-NHL, or HL; only patients with classical HL must have documented histologic demonstration of CD45+ cells adjacent to the Reed Sternberg cells; patients must have received at least one prior standard systemic therapy with documented recurrent or refractory disease; patients with mantle cell lymphoma (MCL), T-NHL, or other high-risk malignancies may be enrolled/transplanted in complete remission (CR)/first partial remission (PR1)
* Creatinine < 2.0
* Bilirubin < 1.5 mg/dL
* All patients eligible for therapeutic study must have a minimum of >= 2 x10^6 CD34/kg autologous hematopoietic stem cells harvested and cryopreserved
* Patients must have an expected survival of > 60 days and must be free of major infection

Exclusion Criteria:

* Circulating human anti-mouse antibody (HAMA), to be determined before each infusion
* Systemic anti-lymphoma therapy given in the previous 30 days before the scheduled therapy dose with the exception of rituximab
* Inability to understand or give an informed consent
* Lymphoma involving the central nervous system
* Other serious medical conditions considered to represent contraindications to ASCT (e.g., abnormally decreased cardiac ejection fraction, diffusion capacity of carbon monoxide [DLCO] < 50% predicted, etc.)
* Known human immunodeficiency virus (HIV) seropositivity
* Pregnancy or breast feeding
* Prior autologous or allogeneic bone marrow or stem cell transplant
* Prior radiation therapy (RT) > 20 gray (Gy) to a critical organ within 1 year of enrollment
* Southwestern Oncology Group (SWOG) performance status >= 2.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10-09 (Actual); Primary Completion 2017-07-26 (Actual); Study Completion 2020-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Gopal, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (90Y-BC8-DOTA, Chemotherapy, PBSC)
Started | 20
Completed | 19
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (90Y-BC8-DOTA, Chemotherapy, PBSC)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum-tolerated Dose (MTD) of Yttrium-90-BC8-DOTA
Description: Single patients will be treated at escalating doses in 2-Gy increments (Table 4) until a DLT is observed. Once a DLT is observed, the second stage will begin at the next lower dose level and patients will be treated in cohorts of 4.
Time Frame: Within 30 days post-transplant
Measure: Number; unit: Gy - MTD
Arm/Group | Treatment (90Y-BC8-DOTA, Chemotherapy, PBSC)
Number analyzed (Participants) | 19
Gy - MTD | 34

2. Primary Outcome: Progression-free Survival Following Autologous Stem Cell Transplant (ASCT)
Description: Estimate the 1 year progression-free survival (PFS) rate after ASCT
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (90Y-BC8-DOTA, Chemotherapy, PBSC)
Number analyzed (Participants) | 19
Participants | 12

3. Secondary Outcome: Estimated Dose to Tumor Sites Based on the Tumor to Normal Organ Ratios Derived From Dosimetry Estimates Coupled With the Absorbed Dose to Normal Organs Based on the Administered Activity of Yttrium Y 90 Anti-CD45 Monoclonal Antibody BC8
Description: Will be evaluated among all patients and among those treated at the estimated MTD.
Time Frame: Up to 5 years
Measure: Number; unit: mCi
Arm/Group | Treatment (90Y-BC8-DOTA, Chemotherapy, PBSC)
Number analyzed (Participants) | 19
mCi | 52.8

4. Secondary Outcome: The Lowest Antibody (Yttrium 90-BC8-DOTA) Dose (mg/kg) That is Consistent With a Favorable Biodistribution Rate >= 80% in Lymphoma Patients
Time Frame: Up to 5 years
Measure: Number; unit: mg/kg
Arm/Group | Treatment (90Y-BC8-DOTA, Chemotherapy, PBSC)
Number analyzed (Participants) | 19
mg/kg | 0.75

ADVERSE EVENTS:
Time Frame: AEs are monitored and recorded from the time of first exposure to the investigational agent (i.e., the start of the 111In-DOTA-BC8 infusion) through day +30 post-transplant or through discharge prior to that date from the SCCA system to care of the patient's primary physician; Beyond day 30 after transplant/discharge from the transplant service until day 100, only SAEs and grade 4 and 5 toxicities will be collected.
Arm/Group | Treatment (90Y-BC8-DOTA, Chemotherapy, PBSC)
All-Cause Mortality (participants affected / at risk) | 5/20
Serious Adverse Events (participants affected / at risk) | 20/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (90Y-BC8-DOTA, Chemotherapy, PBSC) (N=20)
Allergic reaction (Immune system disorders) | 3 (3) — Grade 3
Anaphylaxis (Immune system disorders) | 1 (1) — Grade 3
Anorexia (Metabolism and nutrition disorders) | 5 (5) — Grade 3
Chest pain (Cardiac disorders) | 1 (1) — Grade 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 3
Diarrhea (Gastrointestinal disorders) | 1 (1) — Grade 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 3
Febrile neutropenia (Blood and lymphatic system disorders) | 13 (13) — Grade 3
Fever (General disorders) | 3 (3) — Grade 3
Headache (Nervous system disorders) | 1 (1) — Grade 3
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) — Grade 3
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) — Grade 3
Hypotension (Vascular disorders) | 2 (2) — Grade 2 and Grade 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Grade 3 and Grade 4
Engraftment syndrome (Immune system disorders) | 1 (1) — Grade 3
Blood infection (Infections and infestations) | 2 (2) — Grade 3
Mucositis (Gastrointestinal disorders) | 15 (15) — Grade 3
Nausea (Gastrointestinal disorders) | 2 (2) — Grade 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 3
Peripheral neuropathy (Nervous system disorders) | 1 (1) — Grade 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) — Grade 3
Serum sickness (Immune system disorders) | 2 (2) — Grade 3
Sinusitis (Infections and infestations) | 1 (1) — Grade 3
Syncope (Nervous system disorders) | 2 (2) — Grade 3
Vomiting (Gastrointestinal disorders) | 1 (1) — Grade 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT01921387/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT01921387/SAP_001.pdf